CLINICAL TRIAL: NCT04427995
Title: Standalone OMNI Surgical System for Open-angle Glaucoma
Acronym: OMNIgl
Status: Terminated | Type: Observational
Why Stopped: product expired and could not be resupplied
Sponsor: Iqbal Ahmed (Other)
Collaborators: OMNI Medical Services, LLC (Network)
Responsible Party: Sponsor-Investigator, Iqbal Ahmed, Principal Investigator, Prism Eye Institute
Organization: Prism Eye Institute (Other)
Other Study IDs: 948
Record Dates: First submitted 2020-06-05; First posted 2020-06-11 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Open Angle Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Oen Angle Glaucoma: • Patients aged 30-95 with primary or pigmentary / pseudoexfolliative / juvenile / normal pressure open angle glaucoma or combined mechanism glaucoma with IOP of 10-40 mmHg on maximum tolerated medical therapy who are either progressing, above IOP target, or poorly adherent or tolerant to medical therapy. Phakic or pseudophakic eyes and previous laser trabeculoplasty will be included.
  Interventions: Device: OMNI surgical system

INTERVENTIONS:
Device: OMNI surgical system — GATT + viscodilation
  Other Names: OMNI surgical systems

SUMMARY:
The emergence of minimally invasive glaucoma surgeries (MIGS) has seen a variety of potential innovative surgical alternatives to help better control intraocular pressure (IOP). The OMNI™ Surgical System (Sight Sciences, Menlo Park, CA, USA) is a promising MIGS procedure. It combines two procedures known as trabeculotomy and viscodilation of Schlemm's canal in one hand held device without the need for additional incisions or extra instrumentation. The device recently received FDA approval in the United States for certain indications in ophthalmic surgery. To date, no study has examined the effect of standalone viscodilation and trabeculotomy on glaucoma drop burden and IOP.

DETAILED DESCRIPTION:
The emergence of minimally invasive glaucoma surgeries (MIGS) has seen a variety of potential innovative surgical alternatives to help better control intraocular pressure (IOP).1 The OMNI™ Surgical System (Sight Sciences, Menlo Park, CA, USA) is a promising procedure which targets the conventional outflow pathway.2 This device treats the trabecular meshwork, Schlemm's canal and the distal collector channels, all conventional pathway points of aqueous outflow resistance. Its designed microcatheter allows for cannulation of Schlemm's canal, dilation using the controlled delivery of viscoelastic as well as a trabeculotomy by stripping the trabecular meshwork will retracting the catheter.3 Goniotomy-assisted transluminal trabeculotomy (GATT) has shown promising results in using an ab interno approach to cleave the trabecular meshwork.4 Alternatively, viscodilation alone has also shown an IOP lowering effect. 5 The OMNI Surgical System combines both procedures in one hand held device without the need for additional incisions or extra instrumentation. The device recently received FDA approval in the United States for delivery of small amounts of viscoelastic fluid during ophthalmic surgery and to cut trabecular meshwork tissue during trabeculotomy procedures.6 To date, no study has examined the effect of standalone viscodilation and trabeculotomy on glaucoma drop burden and IOP.

ELIGIBILITY:
Inclusion Criteria

* Patients aged 30-95 with primary or pigmentary / pseudoexfolliative / juvenile / normal pressure open angle glaucoma or combined mechanism glaucoma.
* An IOP of 10-40 mmHg on maximum tolerated medical therapy who are either progressing, above IOP target, or poorly adherent or tolerant to medical therapy.
* Phakic or pseudophakic eyes and previous laser trabeculoplasty will be included.

Exclusion Criteria:

* Other forms of glaucoma,
* prior incisional glaucoma surgery,
* prior corneal graft (PKP, DALK, DSAEK, DMEK),
* Shafer angle grading <2 in 2 or more quadrants.

Ages: 30 Years to 95 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: * Patients aged 30-95 with primary or pigmentary / pseudoexfolliative / juvenile / normal pressure open angle glaucoma or combined mechanism glaucoma with IOP of 10-40 mmHg on maximum tolerated medical therapy who are either progressing, above IOP target, or poorly adherent or tolerant to medical therapy. Phakic or pseudophakic eyes and previous laser trabeculoplasty will be included.
  * Exclusions: Other forms of glaucoma, prior incisional glaucoma surgery, prior corneal graft (PKP, DALK, DSAEK, DMEK), Shafer angle grading <2 in 2 or more quadrants.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Lower Intraocular Pressure and medication dependence | Postoperative week 1, month 1, month 3, annually
  Change in IOP less than or equal to baseline with a medication reduction to 1 or less or an IOP change of 20% or less from baseline with medication

SECONDARY OUTCOMES:
Examine the adverse event profile of the OMNI surgical system in patients with open angle glaucoma. | 1 month post operatively
  Absence of the following complications:
  1. ) Starting after POM1: shallow AC w/ iridocorneal touch, any hyphema, corneal edema, wound leak/dehiscience, choroidal effusion, malignant glaucoma, dellen/non-healing epithelial defect, ptosis, diplopia, and/or; 2.) At any point: additional glaucoma surgery, loss of light perception vision, vitreous hemorrhage, ≥2mm hyphema, hypotony maculopathy, macular edema, choroidal effusion/hemorrhage requiring drainage, suprachoroidal hemorrhage, retinal detachment, endophthalmitis

CONTACTS AND LOCATIONS:
Overall Officials: Iqbal Ahmed, MD, Principal Investigator — Prism Eye Institute
Locations (1):
- Prism Eye Institute, Oakville, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Conlon R, Saheb H, Ahmed II. Glaucoma treatment trends: a review. Can J Ophthalmol. 2017 Feb;52(1):114-124. doi: 10.1016/j.jcjo.2016.07.013. Epub 2016 Nov 17. PMID 28237137
- [Result] Francis BA, Akil H, Bert BB. Ab interno Schlemm's Canal Surgery. Dev Ophthalmol. 2017;59:127-146. doi: 10.1159/000458492. Epub 2017 Apr 25. PMID 28442693
- [Result] Grover DS, Smith O, Fellman RL, Godfrey DG, Gupta A, Montes de Oca I, Feuer WJ. Gonioscopy-assisted Transluminal Trabeculotomy: An Ab Interno Circumferential Trabeculotomy: 24 Months Follow-up. J Glaucoma. 2018 May;27(5):393-401. doi: 10.1097/IJG.0000000000000956. PMID 29613978
- [Result] Gallardo MJ, Supnet RA, Ahmed IIK. Viscodilation of Schlemm's canal for the reduction of IOP via an ab-interno approach. Clin Ophthalmol. 2018 Oct 23;12:2149-2155. doi: 10.2147/OPTH.S177597. eCollection 2018. PMID 30425450
- See also: Related Info — https://omnisurgical.com/.
- See also: Related Info — https://www.accessdata.fda.gov/cdrh_docs/pdf17/K173332.pdf